CLINICAL TRIAL: NCT02414347
Title: F 18 T807 Tau PET Imaging of Alzheimer's Disease [IND# 123119] Protocol A
Brief Title: F 18 T807 Tau PET Imaging of Alzheimer's Disease
Acronym: T807IND
Status: Recruiting | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology & Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IND 123119 Protocol A
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Tauopathies; Brain Diseases; Central Nervous System Diseases; Mild Cognitive Impairment; Nervous System Diseases; Neurodegenerative Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Tauopathies; Brain Diseases; Central Nervous System Diseases; Cognitive Dysfunction; Nervous System Diseases; Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental F 18 T807: Participants will undergo a PET scan using the flortaucipir imaging tracer
  Interventions: Drug: F 18 T807

INTERVENTIONS:
Drug: F 18 T807 — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: 18F-AV-1451

SUMMARY:
A single-center, open-label baseline controlled imaging study designed to assess whether brain tau fibril uptake of flortaucipir as measured by PET correlates with cognitive status of individuals with and without brain tau fibrils.

DETAILED DESCRIPTION:
This project will collect quantitative pilot data that will allow the characterization of uptake and binding of 18F-AV-1451 (also known as F 18 T807), a novel tau imaging compound, in individuals with and without brain tau fibrils. The primary goal is to develop tau imaging technique as an antecedent biomarker of cognitive decline. The investigators propose to obtain preliminary data that will support the possibility of detecting cognitive decline in its earliest stages, before the occurrence of dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, at least 18 years of age.
2. Cognitively normal, or with mild dementia, as assessed clinically
3. Participant is able and willing to undergo testing (MRI or CT, PET, radioactive tracer injection, LP; for those unable to undergo an MRI, CT will be used to generate regions-of-interest).
4. Pre-menopausal women will undergo a urine pregnancy test within 24 hours of drug administration.

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with severe chronic back pain might not be able to lie still during the scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has a high risk for Torsades de Pointes or is taking medications known to prolong QT interval.
4. Has hypersensitivity to F 18 T807 or any of its excipients.
5. Contraindications to PET, PET-CT or MR (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
6. Severe claustrophobia.
7. Currently pregnant or breast-feeding.
8. For those electing to undergo the optional lumbar puncture: currently on anticoagulant of any form -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred (100) participants over a period of approximately 5 years will be enrolled. Participants will undergo an F 18 T807 scan at the Center for Clinical Imaging Research (CCIR) at Washington University using an adaption of the protocol developed by Kolb and colleagues [7]. An MRI may be conducted if one has not been completed within the past 12 months under a related research study.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2014-10-23 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
F 18 T807 Standard Uptake Value Ratios (SUVR) will be correlated with other imaging modalities (MRI, PET amyloid imaging) and cognitive performance. | 5 years
  Employing statistical parametric mapping (SPM), a voxel-based analytic measure in order to quantify and co-localize the imaging patterns from the multiple imaging datasets in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We will share the data with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. We may also share the research data with large data repositories (a repository is a database of information) for broad sharing with the research community. The participant"s individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at this information.

REFERENCES:
- [Background] Day GS, Gordon BA, Perrin RJ, Cairns NJ, Beaumont H, Schwetye K, Ferguson C, Sinha N, Bucelli R, Musiek ES, Ghoshal N, Ponisio MR, Vincent B, Mishra S, Jackson K, Morris JC, Benzinger TLS, Ances BM. In vivo [18F]-AV-1451 tau-PET imaging in sporadic Creutzfeldt-Jakob disease. Neurology. 2018 Mar 6;90(10):e896-e906. doi: 10.1212/WNL.0000000000005064. Epub 2018 Feb 7. PMID 29438042
- [Background] Mishra S, Gordon BA, Su Y, Christensen J, Friedrichsen K, Jackson K, Hornbeck R, Balota DA, Cairns NJ, Morris JC, Ances BM, Benzinger TLS. AV-1451 PET imaging of tau pathology in preclinical Alzheimer disease: Defining a summary measure. Neuroimage. 2017 Nov 1;161:171-178. doi: 10.1016/j.neuroimage.2017.07.050. Epub 2017 Jul 26. PMID 28756238
- [Background] Roe CM, Babulal GM, Mishra S, Gordon BA, Stout SH, Ott BR, Carr DB, Ances BM, Morris JC, Benzinger TLS. Tau and Amyloid Positron Emission Tomography Imaging Predict Driving Performance Among Older Adults with and without Preclinical Alzheimer's Disease. J Alzheimers Dis. 2018;61(2):509-513. doi: 10.3233/JAD-170521. PMID 29171997
- [Background] Gordon BA, McCullough A, Mishra S, Blazey TM, Su Y, Christensen J, Dincer A, Jackson K, Hornbeck RC, Morris JC, Ances BM, Benzinger TLS. Cross-sectional and longitudinal atrophy is preferentially associated with tau rather than amyloid beta positron emission tomography pathology. Alzheimers Dement (Amst). 2018 Mar 6;10:245-252. doi: 10.1016/j.dadm.2018.02.003. eCollection 2018. PMID 29780869
- [Background] Roe CM, Babulal GM, Stout SH, Ott BR, Carr DB, Williams MM, Benzinger TLS, Fagan AM, Holtzman DM, Ances BM, Morris JC. Using the A/T/N Framework to Examine Driving in Preclinical AD. Geriatrics (Basel). 2018 Jun;3(2):23. doi: 10.3390/geriatrics3020023. Epub 2018 May 2. PMID 29805967
- [Background] Strain JF, Smith RX, Beaumont H, Roe CM, Gordon BA, Mishra S, Adeyemo B, Christensen JJ, Su Y, Morris JC, Benzinger TLS, Ances BM. Loss of white matter integrity reflects tau accumulation in Alzheimer disease defined regions. Neurology. 2018 Jul 24;91(4):e313-e318. doi: 10.1212/WNL.0000000000005864. Epub 2018 Jun 29. PMID 29959265
- [Background] Aschenbrenner AJ, Gordon BA, Benzinger TLS, Morris JC, Hassenstab JJ. Influence of tau PET, amyloid PET, and hippocampal volume on cognition in Alzheimer disease. Neurology. 2018 Aug 28;91(9):e859-e866. doi: 10.1212/WNL.0000000000006075. Epub 2018 Aug 1. PMID 30068637
- [Background] Pontecorvo MJ, Devous MD Sr, Navitsky M, Lu M, Salloway S, Schaerf FW, Jennings D, Arora AK, McGeehan A, Lim NC, Xiong H, Joshi AD, Siderowf A, Mintun MA; 18F-AV-1451-A05 investigators. Relationships between flortaucipir PET tau binding and amyloid burden, clinical diagnosis, age and cognition. Brain. 2017 Mar 1;140(3):748-763. doi: 10.1093/brain/aww334. PMID 28077397
- [Background] Zhao Y, Raichle ME, Wen J, Benzinger TL, Fagan AM, Hassenstab J, Vlassenko AG, Luo J, Cairns NJ, Christensen JJ, Morris JC, Yablonskiy DA. In vivo detection of microstructural correlates of brain pathology in preclinical and early Alzheimer Disease with magnetic resonance imaging. Neuroimage. 2017 Mar 1;148:296-304. doi: 10.1016/j.neuroimage.2016.12.026. Epub 2016 Dec 15. PMID 27989773